CLINICAL TRIAL: NCT00778817
Title: Multi-Institutional Phase II Study of IMC-A12, a Recombinant Human IgG1 Monoclonal Antibody Directed at the Type I Insulin-Like Growth Factor Receptor IGF1R, in Adrenocortical Carcinoma: IMC-A12 With Mitotane vs Mitotane Alone
Brief Title: IMC-A12 With Mitotane vs Mitotane Alone in Recurrent, Metastatic, or Primary ACC That Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was permanently halted due to futility concerns.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00291; NCI-2009-00291 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCCRC-16402A; CDR0000617085; 8199 (Other: University of Chicago Comprehensive Cancer Center); 8199 (Other: CTEP); N01CM62201 (NIH); N01CM62205 (NIH); N01CM62204 (NIH); N01CM00100 (NIH); N01CM00038 (NIH); N01CM00099 (NIH); N01CM62207 (NIH); NCT00810537 (obsolete NCT alias)
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Results first posted 2013-11-06 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2013-12

CONDITIONS: Recurrent Adrenocortical Carcinoma; Stage III Adrenocortical Carcinoma; Stage IV Adrenocortical Carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — cixutumumab; Mitotane; Dichlorodiphenyldichloroethane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm II (Mitotane + IMC-A12) (Experimental): Patients receive mitotane as in arm I and anti-IGF-1R recombinant monoclonal antibody IMC-A12 IV over 1 hour once every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: IMC-A12; Drug: mitotane

INTERVENTIONS:
Biological: IMC-A12 — Given IV
  Other Names: anti-IGF-1R recombinant monoclonal antibody IMC-A12; cixutumumab
Drug: mitotane — Given orally
  Other Names: DDD; Lysodren; o,p'-DDD

SUMMARY:
This randomized phase II trial is studying mitotane and IMC-A12 to see how well they work compared with mitotane alone in treating patients with recurrent, metastatic, or primary adrenocortical cancer that cannot be removed by surgery. Drugs used in chemotherapy, such as mitotane, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as IMC-A12, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether mitotane is more effective with or without monoclonal antibody IMC-A12 in treating adrenocortical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the progression-free survival (PFS) rate in patients with recurrent, metastatic, or primary unresectable adrenocortical carcinoma treated with mitotane with vs without anti-IGF-1R recombinant monoclonal antibody IMC-A12 (IMC-A12).

SECONDARY OBJECTIVES:

I. Compare the response rates in these patients using Response Evaluation Criteria in Solid Tumor (RECIST) criteria.

II. Compare the change in tumor size from baseline to 12 weeks in these patients.

III. Compare the overall trajectories in tumor growth in these patients.

TERTIARY OBJECTIVES:

I. Define predictive markers of response or insensitivity to IMC-A12. II. Define pharmacodynamic markers of IMC-A12. III. Determine whether tumor expression of IGF-IR and activation of downstream signaling in archival tumor tissue samples predict efficacy of IMC-A12.

OUTLINE: This is a multicenter study that includes a single-arm safety evaluation phase followed by a randomized phase. Initially, patients are enrolled in the safety evaluation phase. If ≤ 6 of 20 patients experience a dose-limiting toxicity, then the study may proceed to the randomized phase.

SAFETY EVALUATION PHASE: Patients receive oral mitotane once or twice daily and anti-IGF-1R recombinant monoclonal antibody IMC-A12 IV over 1 hour once every 2 weeks in the absence of disease progression or unacceptable toxicity.

RANDOMIZED PHASE: Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral mitotane once or twice daily in the absence of disease progression or unacceptable toxicity. Patients with documented disease progression may cross over and receive treatment on arm II.

ARM II: Patients receive mitotane as in arm I and anti-IGF-1R recombinant monoclonal antibody IMC-A12 IV over 1 hour once every 2 weeks in the absence of disease progression or unacceptable toxicity.

Archival frozen tissue blocks, unstained tumor tissue slides from archival paraffin blocks, plasma samples, and urine samples may be collected and stored for future correlative biomarker studies.

After completion of study therapy, patients are followed up for 6 months.

NOTE: The study was terminated after the safety evaluation phase (i.e., before the randomization phase) due to futility concerns. Thus, patients were only enrolled into ARM II (i.e., mitotate + IMC-A12). Results presented in this report are only given for the safety evaluation phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adrenocortical carcinoma

  * Documented unresectable recurrent, unresectable advanced, or metastatic disease
* At least 1 lesion that can be accurately measured by RECIST criteria as ≥ 20 mm by conventional radiologic techniques or as ≥ 10 mm by spiral CT scan or MRI

  * Patients with disease in an irradiated field as the only site of measurable disease allowed provided there has been a clear progression of the lesion
* No tumors potentially resectable by surgical excision alone
* No known or suspected leptomeningeal disease or brain metastases
* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (transfusion allowed)
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN) OR calculated creatinine clearance ≥ 60 mL/min
* AST or ALT ≤ 3 times ULN
* Total bilirubin ≤ 1.5 times ULN
* HbA1c < 8 within the past 4 weeks
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* Able to take oral medications
* No poor gastrointestinal absorption
* Patients with diabetes mellitus are eligible provided they meet all of the following criteria:

  * Blood glucose is normal (random glucose ≤ 150 mg/dL)
  * HgbA1c ≤ 8 within the past 4 weeks
  * On a stable dietary or therapeutic regimen for the past 2 months
* No active uncontrolled infection
* No severe disease or condition that, in the judgement of the investigator, would make the patient inappropriate for study participation, including, but not limited to:

  * Bleeding diathesis
  * Uncontrolled chronic kidney or liver disease
  * Uncontrolled diabetes
  * History of cardiac history
  * Myocardial infarction within the past 6 months
  * Congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Uncontrolled hypertension
* No current malignancy or previous malignancy with a disease-free interval of < 2 years at the time of diagnosis

  * Patients with adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or skin, or stage A low-grade prostate cancer are eligible
* No known hypersensitivity to monoclonal antibody therapy or mitotane
* No known HIV or hepatitis B or C infection
* No serious medical or psychiatric disorder that would interfere with patient safety or informed consent
* All significant toxic effects of prior surgery resolved to ≤ grade 1 according to NCI CTCAE v. 3.0 criteria
* Mitotane for < 8 weeks prior to study entry AND tolerated it well
* No prior IGFR-directed therapy
* No prior systemic antitumor therapy (cytotoxic chemotherapy, biologic, immunotherapy, or targeted therapy)

  * Prior incomplete surgical resections or radiofrequency ablation or radiotherapy will not be considered as prior therapy provided measurable sites of disease remain
  * Prior adjuvant chemotherapy or mitotane will not be considered as prior antitumor therapy unless it was completed < 6 months before study enrollment
* No prior radiotherapy to > 20% of bone marrow
* More than 4 weeks since prior and no concurrent radiotherapy

  * Radiotherapy for palliation of symptoms related to metastases is permitted provided that it is > 4 weeks from study initiation, and does not involve target/measureable lesions that are followed for drug treatment response evaluation
* No concurrent mitotane ≥ 8 weeks prior to study
* No concurrent tumor resection or tumor-directed surgery
* No other concurrent anticancer or investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2012-05 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hammer, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (8):
- United States (8):
  - University of Southern California, Los Angeles, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Ohio State University Medical Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy and Monoclonal Antibody Therapy: Patients receive mitotane as in arm I and anti-IGF-1R recombinant monoclonal antibody IMC-A12 IV over 1 hour once every 2 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Started | 20
Completed | 16
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate at 6 Weeks
Description: Progression-free survival rates were estimated at 6, 12, and 18 weeks by the Kaplan-Meier method. At a given time point, this outcome is defined as the proportion of subjects who had not progressed or died. Disease progression is defined according to Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0). Progression is characterized by a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 6 weeks
Population: The analysis population excludes two patients who withdrew from the study before the 6 week assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Number analyzed (Participants) | 18
percentage of participants | 50

2. Primary Outcome: Progression-free Survival Rate at 12 Weeks
Description: as for outcome 1
Time Frame: 12 weeks
Population: The analysis population excludes two patients who withdrew from the study before the 6 week assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Number analyzed (Participants) | 18
percentage of participants | 25

3. Primary Outcome: Progression-free Survival Rate at 18 Weeks
Description: as for outcome 1
Time Frame: 18 weeks
Population: The analysis population excludes two patients who withdrew from the study before the 6 week assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Number analyzed (Participants) | 18
percentage of participants | 16.7

4. Secondary Outcome: Best Response Rates
Description: RECIST v1.0 was used to evaluate patient response at each time point. Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter (LD) since the treatment started; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Subjects who were unevaluable for response were classified as having 'Unknown response'.
  Each patient's 'best response' was the most favorable of all recorded responses across all time points. Proportions of patients with each response as their best response are reported in this outcome.
Time Frame: Up to 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Number analyzed (Participants) | 20
percentage of participants
  Progressive disease (PD) | 45
  Stable disease (SD) | 40
  Partial response (PR) | 5
  Complete response (CR) | 0
  Unknown response | 10

5. Secondary Outcome: Response at 6 Weeks
Description: as for outcome 4
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Number analyzed (Participants) | 20
percentage of participants
  Progressive disease (PD) | 45
  Stable disease (SD) | 45
  Partial response (PR) | 0
  Complete response (CR) | 0
  Unknown response | 10

6. Secondary Outcome: Response at 12 Weeks
Description: as for outcome 4
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Number analyzed (Participants) | 20
percentage of participants
  Progressive disease (PD) | 60
  Stable disease (SD) | 30
  Partial response (PR) | 0
  Complete response (CR) | 0
  Unknown response | 10

7. Secondary Outcome: Response at 18 Weeks
Description: as for outcome 4
Time Frame: 18 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Number analyzed (Participants) | 20
percentage of participants
  Progressive disease (PD) | 65
  Stable disease (SD) | 20
  Partial response (PR) | 5
  Complete response (CR) | 0
  Unknown response | 10

8. Secondary Outcome: Response at 48 Weeks
Description: as for outcome 4
Time Frame: 48 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Number analyzed (Participants) | 20
percentage of participants
  Progressive disease (PD) | 65
  Stable disease (SD) | 20
  Partial response (PR) | 5
  Complete response (CR) | 0
  Unknown response | 10

9. Secondary Outcome: Number of Patients Exhibiting Decrease in Tumor Size at 6 Weeks
Description: Total number of patients whose tumor size at 6 weeks was smaller than their tumor size recorded at baseline (by any amount).
Time Frame: 6 weeks
Population: The analysis population excludes two patients who withdrew from the study before the 6 week assessment.
Measure: Number; unit: participants
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Number analyzed (Participants) | 18
participants | 3

10. Secondary Outcome: Number of Patients Exhibiting Decrease in Tumor Size at 12 Weeks
Description: Total number of patients whose tumor size at 12 weeks was smaller than their tumor size recorded at baseline (by any amount).
Time Frame: 12 weeks
Population: The analysis population excludes two patients who withdrew from the study before the 6 week assessment.
Measure: Number; unit: participants
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Number analyzed (Participants) | 18
participants | 3

11. Secondary Outcome: Number of Patients Exhibiting Decrease in Tumor Size at 18 Weeks
Description: Total number of patients whose tumor size at 18 weeks was smaller than their tumor size recorded at baseline (by any amount).
Time Frame: 18 weeks
Population: The analysis population excludes two patients who withdrew from the study before the 6 week assessment.
Measure: Number; unit: participants
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Number analyzed (Participants) | 18
participants | 2

12. Secondary Outcome: Number of Patients Exhibiting Decrease in Tumor Size at 48 Weeks
Description: Total number of patients whose tumor size at 48 weeks was smaller than their tumor size recorded at baseline (by any amount).
Time Frame: 48 weeks
Population: The analysis population excludes two patients who withdrew from the study before the 6 week assessment.
Measure: Number; unit: participants
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Number analyzed (Participants) | 18
participants | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Chemotherapy and Monoclonal Antibody Therapy
Serious Adverse Events (participants affected / at risk) | 9/20
Other Adverse Events (participants affected / at risk) | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy and Monoclonal Antibody Therapy (N=20)
Abdominal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Cholesterol high (Investigations) | 1
Cognitive disturbance (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Multi-organ failure (General disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Tremor (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy and Monoclonal Antibody Therapy (N=20)
Dehydration (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2

LIMITATIONS AND CAVEATS:
After the treatment of 20 subjects, a protocol defined interim analysis was completed for safety and futility. The trial was permanently halted based on futility concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less